CLINICAL TRIAL: NCT05005260
Title: Prospective, Randomized Clinical Trial Comparing Analgesic Efficacy of Liposomal Bupivacaine Single-Injection Interscalene Blockade to Continuous Interscalene Blockade for Patients Undergoing Primary Total Shoulder Arthroplasty
Brief Title: Liposomal Bupivacaine Single-Injection Interscalene Block vs. Continuous Interscalene Block for Primary Total Shoulder Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jason K. Panchamia, D.O., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-000908
Record Dates: First submitted 2021-08-08; First posted 2021-08-13 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Pain, Postoperative; Brachial Plexus Block
Keywords: Interscalene nerve block; total shoulder arthroplasty; pain management; OBAS; QoR-15
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Masking Description: Unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- liposomal bupivacaine single-shot interscalene blockade (Active Comparator): Subjects will receive a preoperative single-injection interscalene nerve block with long-acting numbing medicine, liposomal bupivacaine
  Interventions: Drug: Liposomal bupivacaine + Bupivacaine Hcl 0.5% Inj
- continuous interscalene nerve blockade (Active Comparator): Subjects will receive a preoperative interscalene nerve block with a continuous catheter device which provides local anesthetic, bupivacaine, for up to 3 days.
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: Bupivacaine HCl — Subjects randomized to the continuous interscalene nerve block group will receive a loading dose of 15-20 mL bupivacaine HCl 0.5% followed by a continuous catheter infusion of bupivacaine 0.2% at 8 mL per hour for 72 hours.
  Arms: continuous interscalene nerve blockade
Drug: Liposomal bupivacaine + Bupivacaine Hcl 0.5% Inj — Subjects will receive a one-time interscalene nerve block injection of 5 mL of bupivacaine 0.5% (25 mg) admixed with 10 mL of liposomal bupivacaine (133 mg).
  Arms: liposomal bupivacaine single-shot interscalene blockade

SUMMARY:
This study aims to assess analgesia efficacy between liposomal bupivacaine single injection interscalene blockade vs. continuous interscalene nerve block for patients undergoing primary total shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria

* Adult patients with an American Society of Anesthesiologists (ASA) physiological status I-III
* Patients presenting for unilateral primary total shoulder arthroplasty (includes anatomic and reverse total shoulder arthroplasty).
* Patients 18 years of age and older
* Able to provide informed consent for him or herself

Exclusion Criteria

* Chronic pain syndromes
* Chronic opioid use (>1 month) with OME >5 mg/day OR acute opioid use (< 1 month) with OME > 30 mg/day.
* Body mass index (BMI) > 45 kg/m2
* Severe drug allergy* to medications used in this study, including non-steroidal anti-inflammatory drugs (i.e. celecoxib) and local anesthetics. *defined as an immune reaction resulting in shortness of breath, hives, anaphylaxis, wheezing, and fever
* Personal or family history of malignant hyperthermia.
* Major systemic medical problems such as:

  * Pre-existing severe renal disorder defined as glomerular filtration rate (GFR) <50 units/m2 (if labs are available), currently on dialysis, or highly suspected based on history.
  * Severe hepatic disorder defined as current or past diagnosis of acute/subacute necrosis of liver, acute hepatic failure, chronic liver disease, cirrhosis (primary biliary cirrhosis), chronic hepatitis/toxic hepatitis, liver abscess, hepatic coma, hepatorenal syndrome, other disorders of liver
  * Pre-existing medical history of moderate to severe pulmonary disease requiring medical therapy (obstructive and/or restrictive), use of home oxygen, preoperative baseline oxygen saturation < 93% on room air.
  * History of contralateral hemidiaphragm dysfunction (e.g., paralysis) or phrenic nerve injury.
* Contraindication to a regional anesthesia technique (e.g., preexisting neuropathy+ in the operative extremity, coagulopathy, sepsis, infection at site of injection, uncooperative, and refusal).

  o + pre-existing neuropathy includes sensory and/or motor deficits due to nerve insult of surgical extremity, radicular symptoms of surgical extremity, history of unresolved brachial plexus injury/brachial plexopathy, and tumors of the brachial plexus. Patients with nerve compression distal to site of surgery, such as history of carpal tunnel syndrome or cubital tunnel syndrome, are NOT considered contraindications to regional anesthesia.
* Known to be currently pregnant or actively breastfeeding++

  o ++ All surgical patients are currently screened using a standardized Pregnancy Assessment tool (http://mayoweb.mayo.edu/sp-forms/mc8800-mc8899/mc8801-161.pdf)
* Impaired cognition (e.g. Alzheimer's disease, moderate to severe dementia, encephalopathy)
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason K Panchamia, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine Single-shot Interscalene Blockade | Continuous Interscalene Nerve Blockade
Started | 42 | 46
Completed | 39 | 44
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine Single-shot Interscalene Blockade | Continuous Interscalene Nerve Blockade | Total
Number analyzed (Participants) | 39 | 44 | 83
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [66 to 76] | 69 [66 to 76] | 71 [66 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 22 | 24 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ASA Score [Number; unit: participants] — The American Society of Anesthesiologists (ASA) Physical Status Classification System is a tool used in preparation for surgery to help predict risks in a given patient. The following are classification definitions: ASA 1 - a normal healthy patient, ASA 2 - a patient with mild systemic disease, ASA 3 - a patient with severe systemic disease, ASA 4 - a patient with severe systemic disease that is a constant threat to life, ASA 5 - a moribund patient who is not expected to survive without the operation, ASA 6 - a declared brain-dead patient whose organs are being removed for donor purposes
  participants
    ASA 1 | 1 | 0 | 1
    ASA 2 | 20 | 26 | 46
    ASA 3 | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Score at Rest at 24 Hours Post-operatively
Description: Self-reported pain intensity scores measure using numerical rating scale of 0 (no pain) to 10 (worst pain imaginable). Primary outcome was measured at 24 hours postoperative time point.
Time Frame: Post-Operative Day 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Liposomal Bupivacaine Single-shot Interscalene Blockade | Continuous Interscalene Nerve Blockade
Number analyzed (Participants) | 39 | 44
units on a scale | 1 [0 to 3] | 1 [0 to 2]

2. Secondary Outcome: Cumulative Opioid Consumption
Description: Reported in mg oral morphine equivalents (OME); measured from PACU through postoperative day 3
Time Frame: PACU to postoperative day 3
Measure: Median (Inter-Quartile Range); unit: mg oral morphine equivalents
Arm/Group | Liposomal Bupivacaine Single-shot Interscalene Blockade | Continuous Interscalene Nerve Blockade
Number analyzed (Participants) | 39 | 44
mg oral morphine equivalents | 30.0 [7.5 to 64.0] | 15.0 [7.5 to 38.8]

3. Secondary Outcome: Quality of Recovery Score (QoR)
Description: 15 item short form patient survey using a scoring system evaluating 5 dimensions of health: psychological support, comfort, emotions, physical independence, and pain. The 11-point numerical rating scale leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).
Time Frame: Post-Operative Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine Single-shot Interscalene Blockade | Continuous Interscalene Nerve Blockade
Number analyzed (Participants) | 39 | 44
score on a scale | 126.0 [113.0 to 133.0] | 124.0 [111.0 to 132.5]

ADVERSE EVENTS:
Time Frame: First 3 days after surgery
Arm/Group | Liposomal Bupivacaine Single-shot Interscalene Blockade | Continuous Interscalene Nerve Blockade
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/44
Other Adverse Events (participants affected / at risk) | 0/39 | 7/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Bupivacaine Single-shot Interscalene Blockade (N=39) | Continuous Interscalene Nerve Blockade (N=44)
Leaking catheter (Surgical and medical procedures) | 0 | 5
Catheter dislodgement (Surgical and medical procedures) | 0 | 1
Non-functioning catheter (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT05005260/Prot_SAP_000.pdf